CLINICAL TRIAL: NCT03059992
Title: Open-Label Study to Evaluate the Efficacy and Safety of SCY-078 (Ibrexafungerp) in Patients With Fungal Diseases That Are Refractory to or Intolerant of Standard Antifungal Treatment (FURI)
Brief Title: Study to Evaluate the Efficacy and Safety of Ibrexafungerp in Patients With Fungal Diseases That Are Refractory to or Intolerant of Standard Antifungal Treatment
Acronym: FURI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCY-078-301; 2017-000381-29 (EudraCT Number)
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Invasive Candidiasis; Mucocutaneous Candidiasis; Coccidioidomycosis; Histoplasmosis; Blastomycosis; Chronic Pulmonary Aspergillosis; Allergic Bronchopulmonary Aspergillosis; Invasive Pulmonary Aspergillosis; Recurrent Vulvovaginal Candidiasis; Other Emerging Fungi
MeSH Terms: conditions — Candidiasis, Invasive; Candidiasis, Chronic Mucocutaneous; Coccidioidomycosis; Histoplasmosis; Blastomycosis; Aspergillosis, Allergic Bronchopulmonary; Invasive Pulmonary Aspergillosis; Candidiasis, Vulvovaginal | interventions — ibrexafungerp

STUDY DESIGN:
Intervention Model Description: Open label, non-comparator, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrexafungerp (SCY-078) (Experimental): Ibrexafungerp (SCY-078), 750mg/day orally administered for up to 180 days with loading dose of 1500mg/day (for 2 days) for invasive fungal diseases.
  Interventions: Drug: Ibrexafungerp

INTERVENTIONS:
Drug: Ibrexafungerp — Experimental Study Drug
  Other Names: SCY-078

SUMMARY:
This is a multicenter, open label, non-comparator, single arm study to evaluate the efficacy and safety of ibrexafungerp (SCY-078) in patients ≥ 18 years of age with a documented fungal disease that has been intolerant or refractory (rIFI) to Standard of Care (SoC) antifungal treatment.

DETAILED DESCRIPTION:
This is a multicenter, open label, non-comparator, single arm study to evaluate the efficacy and safety of ibrexafungerp in patients ≥ 18 years of age with a documented invasive and/or severe fungal disease that has been intolerant or refractory (rIFI) to Standard of Care (SoC) antifungal treatment. Patients will be treated with ibrexafungerp for up to 180 days. Treatment beyond 180 days and combination therapy with other antifungal agents may be allowed under special circumstances to be agreed upon by the Investigator and the Sponsor.

Subjects must have a proven or probable fungal disease and meet all study criteria to be considered for enrollment. Eligible subjects must also have documented evidence of failure of, intolerance to, or toxicity related to a currently approved SoC antifungal treatment.

Subjects will also be considered for enrollment if they have an eligible fungal disease and, in the judgement of the investigator, the subject cannot receive approved oral antifungal options (e.g. susceptibility of the organism or risk for drug-drug interactions) and a continued IV antifungal therapy is not desirable or feasible due to clinical or logistical circumstances.

Following a screening visit, there will be up to 15 treatment visits, a follow-up visit and 2 follow-up contacts.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have a documented eligible invasive and/or severe fungal disease that is refractory or intolerant to Standard-of-Care treatment
2. Be able to tolerate medication orally or through a nasogastric (NG) tube or percutaneous endoscopic gastrostomy (PEG) tube
3. Be able to understand and sign a written informed consent form (ICF), which must be obtained prior to treatment and any study-related procedures.
4. Be able to understand and sign a consent or authorization form which shall permit the use, disclosure and transfer of the subject's personal health information. (e.g., in the U.S. HIPAA Authorization form).
5. Be able to understand and follow all study-related procedures including study drug administration.
6. Agree to use a medically acceptable method of contraception while receiving protocol-assigned product.

Key Exclusion Criteria:

1. An invasive fungal disease with CNS involvement.
2. Subject has an inappropriately controlled fungal disease source (e.g., persistent catheters that cannot be removed and are likely the source of infection).
3. Subject is hemodynamically unstable, requiring vasopressor medication for blood pressure support.
4. A life expectancy < 30 days.
5. Subject with abnormal liver test parameters: aspartate aminotransferase (AST), alanine aminotransferase (ALT) >10 x the upper limit of normal (ULN), and/or total bilirubin > 5 x ULN.
6. Subject is pregnant or lactating.
7. Subject has used an investigational drug within 30 days prior to the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis Medical Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Austria (2):
  - Medical University of Graz Department of Internal Medicine, Department of Pulmology, Section for Infectious Disease and Tropical Medicine, Graz
  - Medical University Innsbruck, Innsbruck
- Germany (5):
  - Universitätsklinikum Köln, Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum Essen, Klinik für Infektiologie, Essen
  - Universitätsklinikum Frankfurt, Department of Internal Medicine II, Frankfurt
  - Klinikum St. Georg gGmbH Department for Infectious Disease, Tropical Medicine and Nephrology, Leipzig
  - LMU Klinikum der Universität München, Medizinische Klinik und Poliklinik III, Munich
- Radboud University Medical Center, Department of Medicine Geert Grooteplein Zuid 8, Nijmegen, Gelderland, Netherlands
- Aga Khan University, Karachi, Pakistan
- South Africa (4):
  - Johese Clinical Research, Lyttelton, Centurion
  - Into Research, Groenkloof, Pretoria
  - FCRN Clinical Trial Centre, Three Rivers, Vereeniging
  - Emmed Research, Pretoria
- Spain (2):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - St. George's University of London, London
  - The University of Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis MR, Donnelley MA, Thompson GR. Ibrexafungerp: A novel oral glucan synthase inhibitor. Med Mycol. 2020 Jul 1;58(5):579-592. doi: 10.1093/mmy/myz083. PMID 31342066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibrexafungerp (SCY-078)
Started | 233
Completed | 124
Not Completed | 109

BASELINE CHARACTERISTICS:
Groups:
- Ibrexafungerp (SCY-078): Ibrexafungerp (SCY-078), orally administered QD for up to 180 days.
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (16.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 219
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 180
  More than one race | 1
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a Global Response as Determined by the Data Review Committee (DRC) by Fungal Disease.
Description: The percentage of participants who achieve Global Response (defined as complete or partial response) as determined by the DRC at disease specific timepoints by fungal disease. Global Response is measured by participant survival and overall effect of treatment on the disease. Complete response: Survival, all attributable signs/symptoms (including radiological) resolved and myoclogical eradication of disease; Partial response: Survival, improvement of attributable signs/symptoms (including radiological).
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases.
Time Frame: Vulvovaginal Candidiasis: Day 17. Chronic Mucocutaneous Candidiasis: EOT up to Day 84. Chronic Pulmonary Aspergillus and Allergic Bronchopulmonary Aspergillosis: EOT up to Day 90. All other diseases: EOT up to Day 180. All Days measured from Baseline.
Population: Intent to Treat (ITT) Population - all participants who were enrolled in the study and received at least one dose of study drug.
  Per Protocol (PP) Population - include all ITT participants who received enough study drug to enable clinical efficacy judgement as determined by the DRC, who have an EOT or TOC (as applicable) assessment and who have no major protocol violations that could impact the assessment of efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Overall Study (ITT): Success | 142
  Overall Study (ITT): Failure | 69
  Overall Study (ITT): Not Evaluable | 22
  Overall Study (PP): number analyzed (Participants) | 195
  Overall Study (PP): Success | 131
  Overall Study (PP): Failure | 59
  Overall Study (PP): Not Evaluable | 5
  Acute Invasive Candidiasis including Candidemia (ITT): number analyzed (Participants) | 61
  Acute Invasive Candidiasis including Candidemia (ITT): Success | 40
  Acute Invasive Candidiasis including Candidemia (ITT): Failure | 13
  Acute Invasive Candidiasis including Candidemia (ITT): Not Evaluable | 8
  Acute Invasive Candidiasis including Candidemia (PP): number analyzed (Participants) | 49
  Acute Invasive Candidiasis including Candidemia (PP): Success | 37
  Acute Invasive Candidiasis including Candidemia (PP): Failure | 10
  Acute Invasive Candidiasis including Candidemia (PP): Not Evaluable | 2
  Chronic Invasive Candidiasis (ITT): number analyzed (Participants) | 43
  Chronic Invasive Candidiasis (ITT): Success | 30
  Chronic Invasive Candidiasis (ITT): Failure | 9
  Chronic Invasive Candidiasis (ITT): Not Evaluable | 4
  Chronic Invasive Candidiasis (PP): number analyzed (Participants) | 33
  Chronic Invasive Candidiasis (PP): Success | 25
  Chronic Invasive Candidiasis (PP): Failure | 7
  Chronic Invasive Candidiasis (PP): Not Evaluable | 1
  Esophageal Candidiasis (ITT): number analyzed (Participants) | 16
  Esophageal Candidiasis (ITT): Success | 9
  Esophageal Candidiasis (ITT): Failure | 5
  Esophageal Candidiasis (ITT): Not Evaluable | 2
  Esophageal Candidiasis (PP): number analyzed (Participants) | 14
  Esophageal Candidiasis (PP): Success | 9
  Esophageal Candidiasis (PP): Failure | 4
  Esophageal Candidiasis (PP): Not Evaluable | 1
  Oropharyngeal Candidiasis (ITT): number analyzed (Participants) | 14
  Oropharyngeal Candidiasis (ITT): Success | 9
  Oropharyngeal Candidiasis (ITT): Failure | 5
  Oropharyngeal Candidiasis (ITT): Not Evaluable | 0
  Oropharyngeal Candidiasis (PP): number analyzed (Participants) | 13
  Oropharyngeal Candidiasis (PP): Success | 8
  Oropharyngeal Candidiasis (PP): Failure | 5
  Oropharyngeal Candidiasis (PP): Not Evaluable | 0
  Chronic Mucocutaneous Candidiasis (ITT): number analyzed (Participants) | 13
  Chronic Mucocutaneous Candidiasis (ITT): Success | 8
  Chronic Mucocutaneous Candidiasis (ITT): Failure | 5
  Chronic Mucocutaneous Candidiasis (ITT): Not Evaluable | 0
  Chronic Mucocutaneous Candidiasis (PP): number analyzed (Participants) | 12
  Chronic Mucocutaneous Candidiasis (PP): Success | 8
  Chronic Mucocutaneous Candidiasis (PP): Failure | 4
  Chronic Mucocutaneous Candidiasis (PP): Not Evaluable | 0
  Vulvovaginal Candidiasis (ITT): number analyzed (Participants) | 32
  Vulvovaginal Candidiasis (ITT): Success | 26
  Vulvovaginal Candidiasis (ITT): Failure | 4
  Vulvovaginal Candidiasis (ITT): Not Evaluable | 2
  Vulvovaginal Candidiasis (PP): number analyzed (Participants) | 27
  Vulvovaginal Candidiasis (PP): Success | 24
  Vulvovaginal Candidiasis (PP): Failure | 3
  Vulvovaginal Candidiasis (PP): Not Evaluable | 0
  Disseminated/Invasive Dimorphic Fungi (ITT): number analyzed (Participants) | 3
  Disseminated/Invasive Dimorphic Fungi (ITT): Success | 1
  Disseminated/Invasive Dimorphic Fungi (ITT): Failure | 2
  Disseminated/Invasive Dimorphic Fungi (ITT): Not Evaluable | 0
  Disseminated/Invasive Dimorphic Fungi (PP): number analyzed (Participants) | 3
  Disseminated/Invasive Dimorphic Fungi (PP): Success | 1
  Disseminated/Invasive Dimorphic Fungi (PP): Failure | 2
  Disseminated/Invasive Dimorphic Fungi (PP): Not Evaluable | 0
  Chronic Pulmonary Aspergillosis (ITT): number analyzed (Participants) | 6
  Chronic Pulmonary Aspergillosis (ITT): Success | 0
  Chronic Pulmonary Aspergillosis (ITT): Failure | 6
  Chronic Pulmonary Aspergillosis (ITT): Not Evaluable | 0
  Chronic Pulmonary Aspergillosis (PP): number analyzed (Participants) | 5
  Chronic Pulmonary Aspergillosis (PP): Success | 0
  Chronic Pulmonary Aspergillosis (PP): Failure | 5
  Chronic Pulmonary Aspergillosis (PP): Not Evaluable | 0
  Allergic Bronchopulmonary Aspergillosis (ITT): number analyzed (Participants) | 5
  Allergic Bronchopulmonary Aspergillosis (ITT): Success | 0
  Allergic Bronchopulmonary Aspergillosis (ITT): Failure | 3
  Allergic Bronchopulmonary Aspergillosis (ITT): Not Evaluable | 2
  Allergic Bronchopulmonary Aspergillosis (PP): number analyzed (Participants) | 3
  Allergic Bronchopulmonary Aspergillosis (PP): Success | 0
  Allergic Bronchopulmonary Aspergillosis (PP): Failure | 3
  Allergic Bronchopulmonary Aspergillosis (PP): Not Evaluable | 0
  Invasive Pulmonary Aspergillosis (ITT): number analyzed (Participants) | 29
  Invasive Pulmonary Aspergillosis (ITT): Success | 12
  Invasive Pulmonary Aspergillosis (ITT): Failure | 14
  Invasive Pulmonary Aspergillosis (ITT): Not Evaluable | 3
  Invasive Pulmonary Aspergillosis (PP): number analyzed (Participants) | 26
  Invasive Pulmonary Aspergillosis (PP): Success | 12
  Invasive Pulmonary Aspergillosis (PP): Failure | 13
  Invasive Pulmonary Aspergillosis (PP): Not Evaluable | 1
  Other Emerging Fungi (ITT): number analyzed (Participants) | 11
  Other Emerging Fungi (ITT): Success | 7
  Other Emerging Fungi (ITT): Failure | 3
  Other Emerging Fungi (ITT): Not Evaluable | 1
  Other Emerging Fungi (PP): number analyzed (Participants) | 10
  Other Emerging Fungi (PP): Success | 7
  Other Emerging Fungi (PP): Failure | 3
  Other Emerging Fungi (PP): Not Evaluable | 0

2. Secondary Outcome: Percentage of Participants Who Achieve a Global Response as Determined by the Data Review Committee (DRC) by Enrollment Category
Description: The percentage of participants who achieve a Global Response (defined as complete or partial response) as determined by the DRC by enrollment category, at disease specific timepoints. Global Response is measured by participant survival and overall effect of treatment on the disease. Complete response: Survival, all attributable signs/symptoms (including radiological) resolved and myoclogical eradication of disease; Partial response: Survival, improvement of attributable signs/symptoms (including radiological).
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Participants may have been enrolled for more than 1 enrollment reason.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) Population - all participants who were enrolled in the study and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Refractory Fungal Infection: number analyzed (Participants) | 128
  Refractory Fungal Infection: Success | 74
  Refractory Fungal Infection: Failure | 41
  Refractory Fungal Infection: Not Evaluable | 13
  Resistance to standard of care antifungal: number analyzed (Participants) | 134
  Resistance to standard of care antifungal: Success | 95
  Resistance to standard of care antifungal: Failure | 29
  Resistance to standard of care antifungal: Not Evaluable | 10
  Intolerance to standard of care antifungal: number analyzed (Participants) | 29
  Intolerance to standard of care antifungal: Success | 13
  Intolerance to standard of care antifungal: Failure | 14
  Intolerance to standard of care antifungal: Not Evaluable | 2
  Toxicities associated with standard of care antifungal: number analyzed (Participants) | 17
  Toxicities associated with standard of care antifungal: Success | 7
  Toxicities associated with standard of care antifungal: Failure | 8
  Toxicities associated with standard of care antifungal: Not Evaluable | 2
  Relapse: number analyzed (Participants) | 18
  Relapse: Success | 12
  Relapse: Failure | 5
  Relapse: Not Evaluable | 1
  Other: number analyzed (Participants) | 2
  Other: Success | 0
  Other: Failure | 1
  Other: Not Evaluable | 1

3. Secondary Outcome: Percentage of Participants Who Achieve a Global Response as Determined by the Data Review Committee (DRC) by Disease Category.
Description: The percentage of participants who achieve Global Response (defined as complete or partial response) as determined by the DRC at disease specific timepoints by disease category. Global Response is measured by participant survival and overall effect of treatment on the disease. Complete response: Survival, all attributable signs/symptoms (including radiological) resolved and myoclogical eradication of disease; Partial response: Survival, improvement of attributable signs/symptoms (including radiological).
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Invasive Candidiasis including Candidemia: number analyzed (Participants) | 104
  Invasive Candidiasis including Candidemia: Success | 70
  Invasive Candidiasis including Candidemia: Failure | 22
  Invasive Candidiasis including Candidemia: Not Evaluable | 12
  Mucocutaneous Candidiasis: number analyzed (Participants) | 75
  Mucocutaneous Candidiasis: Success | 52
  Mucocutaneous Candidiasis: Failure | 19
  Mucocutaneous Candidiasis: Not Evaluable | 4
  Dimorphic Fungi: number analyzed (Participants) | 3
  Dimorphic Fungi: Success | 1
  Dimorphic Fungi: Failure | 2
  Dimorphic Fungi: Not Evaluable | 0
  Aspergillus Syndromes: number analyzed (Participants) | 40
  Aspergillus Syndromes: Success | 12
  Aspergillus Syndromes: Failure | 23
  Aspergillus Syndromes: Not Evaluable | 5
  Other emerging fungi: number analyzed (Participants) | 11
  Other emerging fungi: Success | 7
  Other emerging fungi: Failure | 3
  Other emerging fungi: Not Evaluable | 1

4. Secondary Outcome: Percentage of Participants With a Clinical Response (Based on Signs and Symptoms) by Disease Category
Description: The percentage of participants with a Clinical Response as determined by the DRC at disease specific timepoints, by disease category. Clinical Response: resolution or improvement in attributable symptoms and signs of disease and radiological abnormalities (if applicable) .
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Clinical response was evaluated based on disease signs (including radiological signs) and symptoms.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Invasive Candidiasis including Candidemia: number analyzed (Participants) | 104
  Invasive Candidiasis including Candidemia: Success | 57
  Invasive Candidiasis including Candidemia: Failure | 16
  Invasive Candidiasis including Candidemia: Not Evaluable | 29
  Invasive Candidiasis including Candidemia: No Response | 2
  Mucocutaneous Candidiasis (TOC): number analyzed (Participants) | 75
  Mucocutaneous Candidiasis (TOC): Success | 25
  Mucocutaneous Candidiasis (TOC): Failure | 5
  Mucocutaneous Candidiasis (TOC): Not Evaluable | 2
  Mucocutaneous Candidiasis (TOC): No Response | 43
  Dimorphic Fungi: number analyzed (Participants) | 3
  Dimorphic Fungi: Success | 3
  Dimorphic Fungi: Failure | 0
  Dimorphic Fungi: Not Evaluable | 0
  Dimorphic Fungi: No Response | 0
  Aspergillus Syndromes: number analyzed (Participants) | 40
  Aspergillus Syndromes: Success | 18
  Aspergillus Syndromes: Failure | 14
  Aspergillus Syndromes: Not Evaluable | 6
  Aspergillus Syndromes: No Response | 2
  Other emerging fungi: number analyzed (Participants) | 11
  Other emerging fungi: Success | 7
  Other emerging fungi: Failure | 3
  Other emerging fungi: Not Evaluable | 1
  Other emerging fungi: No Response | 0

5. Secondary Outcome: Percentage of Participants With a Clinical Response (Signs and Symptoms) by Disease Category and Pathogen
Description: The percentage of participants with a Clinical Response as determined by the DRC by disease category and by pathogen isolated, at disease specific timepoints. Clinical Response: resolution or improvement in attributable symptoms and signs of disease and radiological abnormalities (if applicable) .
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Clinical response was evaluated based on disease signs (including radiological signs) and symptoms.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Invasive Candidiasis, including Candidemia (C. albicans): number analyzed (Participants) | 26
  Invasive Candidiasis, including Candidemia (C. albicans): Success | 11
  Invasive Candidiasis, including Candidemia (C. albicans): Failure | 7
  Invasive Candidiasis, including Candidemia (C. albicans): Not Evaluable/Missing | 8
  Invasive Candidiasis, including Candidemia (C. auris): number analyzed (Participants) | 10
  Invasive Candidiasis, including Candidemia (C. auris): Success | 6
  Invasive Candidiasis, including Candidemia (C. auris): Failure | 1
  Invasive Candidiasis, including Candidemia (C. auris): Not Evaluable/Missing | 3
  Invasive Candidiasis, including Candidemia (C. glabrata): number analyzed (Participants) | 49
  Invasive Candidiasis, including Candidemia (C. glabrata): Success | 30
  Invasive Candidiasis, including Candidemia (C. glabrata): Failure | 6
  Invasive Candidiasis, including Candidemia (C. glabrata): Not Evaluable/Missing | 13
  Invasive Candidiasis, including Candidemia (C. krusei): number analyzed (Participants) | 8
  Invasive Candidiasis, including Candidemia (C. krusei): Success | 4
  Invasive Candidiasis, including Candidemia (C. krusei): Failure | 2
  Invasive Candidiasis, including Candidemia (C. krusei): Not Evaluable/Missing | 2
  Invasive Candidiasis, including Candidemia (C. parapsilosis): number analyzed (Participants) | 9
  Invasive Candidiasis, including Candidemia (C. parapsilosis): Success | 5
  Invasive Candidiasis, including Candidemia (C. parapsilosis): Failure | 1
  Invasive Candidiasis, including Candidemia (C. parapsilosis): Not Evaluable/Missing | 3
  Invasive Candidiasis, including Candidemia (C. tropicalis): number analyzed (Participants) | 9
  Invasive Candidiasis, including Candidemia (C. tropicalis): Success | 6
  Invasive Candidiasis, including Candidemia (C. tropicalis): Failure | 0
  Invasive Candidiasis, including Candidemia (C. tropicalis): Not Evaluable/Missing | 3
  Invasive Candidiasis, including Candidemia (other): number analyzed (Participants) | 5
  Invasive Candidiasis, including Candidemia (other): Success | 3
  Invasive Candidiasis, including Candidemia (other): Failure | 0
  Invasive Candidiasis, including Candidemia (other): Not Evaluable/Missing | 2
  Mucocutaneous Candidiasis (C. albicans): number analyzed (Participants) | 47
  Mucocutaneous Candidiasis (C. albicans): Success | 19
  Mucocutaneous Candidiasis (C. albicans): Failure | 1
  Mucocutaneous Candidiasis (C. albicans): Not Evaluable/Missing | 27
  Mucocutaneous Candidiasis (C. glabrata): number analyzed (Participants) | 25
  Mucocutaneous Candidiasis (C. glabrata): Success | 5
  Mucocutaneous Candidiasis (C. glabrata): Failure | 3
  Mucocutaneous Candidiasis (C. glabrata): Not Evaluable/Missing | 17
  Mucocutaneous Candidiasis (C. krusei): number analyzed (Participants) | 7
  Mucocutaneous Candidiasis (C. krusei): Success | 2
  Mucocutaneous Candidiasis (C. krusei): Failure | 1
  Mucocutaneous Candidiasis (C. krusei): Not Evaluable/Missing | 4
  Mucocutaneous Candidiasis (C. tropicalis): number analyzed (Participants) | 1
  Mucocutaneous Candidiasis (C. tropicalis): Success | 0
  Mucocutaneous Candidiasis (C. tropicalis): Failure | 0
  Mucocutaneous Candidiasis (C. tropicalis): Not Evaluable/Missing | 1
  Mucocutaneous Candidiasis (C. parapsilosis): number analyzed (Participants) | 1
  Mucocutaneous Candidiasis (C. parapsilosis): Success | 1
  Mucocutaneous Candidiasis (C. parapsilosis): Failure | 0
  Mucocutaneous Candidiasis (C. parapsilosis): Not Evaluable/Missing | 0
  Mucocutaneous Candidiasis (other): number analyzed (Participants) | 9
  Mucocutaneous Candidiasis (other): Success | 3
  Mucocutaneous Candidiasis (other): Failure | 1
  Mucocutaneous Candidiasis (other): Not Evaluable/Missing | 5
  Dimorphic Fungi (Histoplasmosis): number analyzed (Participants) | 3
  Dimorphic Fungi (Histoplasmosis): Success | 3
  Dimorphic Fungi (Histoplasmosis): Failure | 0
  Dimorphic Fungi (Histoplasmosis): Not Evaluable/Missing | 0
  Aspergillus Syndromes (A. flavus): number analyzed (Participants) | 2
  Aspergillus Syndromes (A. flavus): Success | 2
  Aspergillus Syndromes (A. flavus): Failure | 0
  Aspergillus Syndromes (A. flavus): Not Evaluable/Missing | 0
  Aspergillus Syndromes (A. fumigatus): number analyzed (Participants) | 18
  Aspergillus Syndromes (A. fumigatus): Success | 8
  Aspergillus Syndromes (A. fumigatus): Failure | 8
  Aspergillus Syndromes (A. fumigatus): Not Evaluable/Missing | 2
  Aspergillus Syndromes (other): number analyzed (Participants) | 14
  Aspergillus Syndromes (other): Success | 9
  Aspergillus Syndromes (other): Failure | 5
  Aspergillus Syndromes (other): Not Evaluable/Missing | 0

6. Secondary Outcome: Percentage of Participants With a Clinical Response (Signs and Symptoms) by Fungal Disease
Description: The percentage of participants with a Clinical Response as determined by the DRC by fungal disease, at disease specific timepoints. Clinical Response: resolution or improvement in attributable symptoms and signs of disease and radiological abnormalities (if applicable) .
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Clinical response was evaluated based on disease signs (including radiological signs) and symptoms.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Acute Invasive Candidiasis, including Candidemia: number analyzed (Participants) | 61
  Acute Invasive Candidiasis, including Candidemia: Success | 30
  Acute Invasive Candidiasis, including Candidemia: Failure | 10
  Acute Invasive Candidiasis, including Candidemia: Not Evaluable | 19
  Acute Invasive Candidiasis, including Candidemia: No Response | 2
  Chronic Invasive Candidiasis: number analyzed (Participants) | 43
  Chronic Invasive Candidiasis: Success | 27
  Chronic Invasive Candidiasis: Failure | 6
  Chronic Invasive Candidiasis: Not Evaluable | 10
  Chronic Invasive Candidiasis: No Response | 0
  Vulvovaginal Candidiasis: number analyzed (Participants) | 32
  Vulvovaginal Candidiasis: Success | 25
  Vulvovaginal Candidiasis: Failure | 5
  Vulvovaginal Candidiasis: Not Evaluable | 2
  Vulvovaginal Candidiasis: No Response | 0
  Esophageal Candidiasis: number analyzed (Participants) | 16
  Esophageal Candidiasis: Success | 10
  Esophageal Candidiasis: Failure | 4
  Esophageal Candidiasis: Not Evaluable | 2
  Esophageal Candidiasis: No Response | 0
  Oropharyngeal Candidiasis: number analyzed (Participants) | 14
  Oropharyngeal Candidiasis: Success | 10
  Oropharyngeal Candidiasis: Failure | 4
  Oropharyngeal Candidiasis: Not Evaluable | 0
  Oropharyngeal Candidiasis: No Response | 0
  Chronic Mucocutaneous Candidiasis: number analyzed (Participants) | 13
  Chronic Mucocutaneous Candidiasis: Success | 8
  Chronic Mucocutaneous Candidiasis: Failure | 5
  Chronic Mucocutaneous Candidiasis: Not Evaluable | 0
  Chronic Mucocutaneous Candidiasis: No Response | 0
  Disseminated/Invasive Dimorphic Fungi: number analyzed (Participants) | 3
  Disseminated/Invasive Dimorphic Fungi: Success | 3
  Disseminated/Invasive Dimorphic Fungi: Failure | 0
  Disseminated/Invasive Dimorphic Fungi: Not Evaluable | 0
  Disseminated/Invasive Dimorphic Fungi: No Response | 0
  Chronic Pulmonary Aspergillosis: number analyzed (Participants) | 6
  Chronic Pulmonary Aspergillosis: Success | 3
  Chronic Pulmonary Aspergillosis: Failure | 2
  Chronic Pulmonary Aspergillosis: Not Evaluable | 1
  Chronic Pulmonary Aspergillosis: No Response | 0
  Allergic Bronchopulmonary Aspergillosis: number analyzed (Participants) | 5
  Allergic Bronchopulmonary Aspergillosis: Success | 0
  Allergic Bronchopulmonary Aspergillosis: Failure | 2
  Allergic Bronchopulmonary Aspergillosis: Not Evaluable | 2
  Allergic Bronchopulmonary Aspergillosis: No Response | 1
  Invasive Pulmonary Aspergillosis: number analyzed (Participants) | 29
  Invasive Pulmonary Aspergillosis: Success | 15
  Invasive Pulmonary Aspergillosis: Failure | 10
  Invasive Pulmonary Aspergillosis: Not Evaluable | 3
  Invasive Pulmonary Aspergillosis: No Response | 1
  Other Emerging Fungi: number analyzed (Participants) | 11
  Other Emerging Fungi: Success | 7
  Other Emerging Fungi: Failure | 3
  Other Emerging Fungi: Not Evaluable | 1
  Other Emerging Fungi: No Response | 0

7. Secondary Outcome: Percentage of Participants With a Clinical Response (Signs and Symptoms) by Enrollment Category
Description: The percentage of participants with a Clinical Response as determined by the DRC by enrollment category, at disease specific timepoints. Clinical Response: resolution or improvement in attributable symptoms and signs of disease and radiological abnormalities (if applicable) .
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Clinical response was evaluated based on disease signs (including radiological signs) and symptoms.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Refractory: number analyzed (Participants) | 128
  Refractory: Success | 57
  Refractory: Failure | 29
  Refractory: Not Evaluable | 13
  Refractory: No Response | 29
  Resistence: number analyzed (Participants) | 134
  Resistence: Success | 75
  Resistence: Failure | 23
  Resistence: Not Evaluable | 25
  Resistence: No Response | 11
  Intolerance: number analyzed (Participants) | 29
  Intolerance: Success | 16
  Intolerance: Failure | 8
  Intolerance: Not Evaluable | 3
  Intolerance: No Response | 2
  Toxicities: number analyzed (Participants) | 17
  Toxicities: Success | 12
  Toxicities: Failure | 3
  Toxicities: Not Evaluable | 1
  Toxicities: No Response | 1
  Relapse: number analyzed (Participants) | 18
  Relapse: Success | 8
  Relapse: Failure | 4
  Relapse: Not Evaluable | 1
  Relapse: No Response | 5

8. Secondary Outcome: Percentage of Participants With a Mycological Response by Disease Category
Description: The percentage of participants with a Mycological Response as determined by the DRC by disease category, at disease specific timepoints. Mycological Response: evidence of eradication or clearance of cultures or reduction of fungal burden, as assessed by a quantitative and validated laboratory marker.
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Mycological response was evaluated based on culture, microscopy and other biomarkers of fungal infection.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Invasive Candidiasis including Candidemia: number analyzed (Participants) | 104
  Invasive Candidiasis including Candidemia: Success | 20
  Invasive Candidiasis including Candidemia: Failure | 14
  Invasive Candidiasis including Candidemia: Not Evaluable/Missing | 70
  Mucocutaneous Candidiasis (TOC): number analyzed (Participants) | 75
  Mucocutaneous Candidiasis (TOC): Success | 11
  Mucocutaneous Candidiasis (TOC): Failure | 13
  Mucocutaneous Candidiasis (TOC): Not Evaluable/Missing | 51
  Dimorphic Fungi: number analyzed (Participants) | 3
  Dimorphic Fungi: Success | 0
  Dimorphic Fungi: Failure | 1
  Dimorphic Fungi: Not Evaluable/Missing | 2
  Aspergillus Syndromes: number analyzed (Participants) | 40
  Aspergillus Syndromes: Success | 5
  Aspergillus Syndromes: Failure | 13
  Aspergillus Syndromes: Not Evaluable/Missing | 22
  Other emerging fungi: number analyzed (Participants) | 11
  Other emerging fungi: Success | 2
  Other emerging fungi: Failure | 2
  Other emerging fungi: Not Evaluable/Missing | 7

9. Secondary Outcome: Percentage of Participants With a Mycological Response by Disease Category and Pathogen
Description: The percentage of participants with a Mycological Response as determined by the DRC by disease category and by pathogen, at disease specific timepoints. Mycological Response: evidence of eradication or clearance of cultures or reduction of fungal burden, as assessed by a quantitative and validated laboratory marker.
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Mycological response was evaluated based on culture, microscopy and other biomarkers of fungal infection.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Invasive Candidiasis, including Candidemia (C. albicans): number analyzed (Participants) | 26
  Invasive Candidiasis, including Candidemia (C. albicans): Success | 3
  Invasive Candidiasis, including Candidemia (C. albicans): Failure | 6
  Invasive Candidiasis, including Candidemia (C. albicans): Not Evaluable/Missing | 17
  Invasive Candidiasis, including Candidemia (C. parapsilosis): number analyzed (Participants) | 9
  Invasive Candidiasis, including Candidemia (C. parapsilosis): Success | 1
  Invasive Candidiasis, including Candidemia (C. parapsilosis): Failure | 2
  Invasive Candidiasis, including Candidemia (C. parapsilosis): Not Evaluable/Missing | 6
  Invasive Candidiasis, including Candidemia (C. auris): number analyzed (Participants) | 10
  Invasive Candidiasis, including Candidemia (C. auris): Success | 2
  Invasive Candidiasis, including Candidemia (C. auris): Failure | 1
  Invasive Candidiasis, including Candidemia (C. auris): Not Evaluable/Missing | 7
  Invasive Candidiasis, including Candidemia (C. glabrata): number analyzed (Participants) | 49
  Invasive Candidiasis, including Candidemia (C. glabrata): Success | 10
  Invasive Candidiasis, including Candidemia (C. glabrata): Failure | 7
  Invasive Candidiasis, including Candidemia (C. glabrata): Not Evaluable/Missing | 32
  Invasive Candidiasis, including Candidemia (C. krusei): number analyzed (Participants) | 8
  Invasive Candidiasis, including Candidemia (C. krusei): Success | 5
  Invasive Candidiasis, including Candidemia (C. krusei): Failure | 0
  Invasive Candidiasis, including Candidemia (C. krusei): Not Evaluable/Missing | 3
  Invasive Candidiasis, including Candidemia (C. tropicalis): number analyzed (Participants) | 9
  Invasive Candidiasis, including Candidemia (C. tropicalis): Success | 2
  Invasive Candidiasis, including Candidemia (C. tropicalis): Failure | 0
  Invasive Candidiasis, including Candidemia (C. tropicalis): Not Evaluable/Missing | 7
  Invasive Candidiasis, including Candidemia (other): number analyzed (Participants) | 5
  Invasive Candidiasis, including Candidemia (other): Success | 0
  Invasive Candidiasis, including Candidemia (other): Failure | 0
  Invasive Candidiasis, including Candidemia (other): Not Evaluable/Missing | 5
  Mucocutaneous Candidiasis (C. albicans): number analyzed (Participants) | 47
  Mucocutaneous Candidiasis (C. albicans): Success | 10
  Mucocutaneous Candidiasis (C. albicans): Failure | 5
  Mucocutaneous Candidiasis (C. albicans): Not Evaluable/Missing | 32
  Mucocutaneous Candidiasis (C. glabrata): number analyzed (Participants) | 25
  Mucocutaneous Candidiasis (C. glabrata): Success | 0
  Mucocutaneous Candidiasis (C. glabrata): Failure | 8
  Mucocutaneous Candidiasis (C. glabrata): Not Evaluable/Missing | 17
  Mucocutaneous Candidiasis (C. krusei): number analyzed (Participants) | 7
  Mucocutaneous Candidiasis (C. krusei): Success | 2
  Mucocutaneous Candidiasis (C. krusei): Failure | 1
  Mucocutaneous Candidiasis (C. krusei): Not Evaluable/Missing | 4
  Mucocutaneous Candidiasis (C. parapsilosis): number analyzed (Participants) | 1
  Mucocutaneous Candidiasis (C. parapsilosis): Success | 0
  Mucocutaneous Candidiasis (C. parapsilosis): Failure | 0
  Mucocutaneous Candidiasis (C. parapsilosis): Not Evaluable/Missing | 1
  Mucocutaneous Candidiasis (C. tropicalis): number analyzed (Participants) | 1
  Mucocutaneous Candidiasis (C. tropicalis): Success | 0
  Mucocutaneous Candidiasis (C. tropicalis): Failure | 0
  Mucocutaneous Candidiasis (C. tropicalis): Not Evaluable/Missing | 1
  Mucocutaneous Candidiasis other): number analyzed (Participants) | 9
  Mucocutaneous Candidiasis other): Success | 2
  Mucocutaneous Candidiasis other): Failure | 2
  Mucocutaneous Candidiasis other): Not Evaluable/Missing | 5
  Dimorphic Fungi (Coccidioidomycosis): number analyzed (Participants) | 0
  Dimorphic Fungi (Coccidioidomycosis): Success | 0
  Dimorphic Fungi (Coccidioidomycosis): Failure | 0
  Dimorphic Fungi (Coccidioidomycosis): Not Evaluable/Missing | 0
  Dimorphic Fungi (Histoplasmosis): number analyzed (Participants) | 3
  Dimorphic Fungi (Histoplasmosis): Success | 0
  Dimorphic Fungi (Histoplasmosis): Failure | 1
  Dimorphic Fungi (Histoplasmosis): Not Evaluable/Missing | 2
  Aspergillus Syndromes (A. nidulans): number analyzed (Participants) | 1
  Aspergillus Syndromes (A. nidulans): Success | 0
  Aspergillus Syndromes (A. nidulans): Failure | 1
  Aspergillus Syndromes (A. nidulans): Not Evaluable/Missing | 0
  Aspergillus Syndromes (A. fumigatus): number analyzed (Participants) | 18
  Aspergillus Syndromes (A. fumigatus): Success | 1
  Aspergillus Syndromes (A. fumigatus): Failure | 5
  Aspergillus Syndromes (A. fumigatus): Not Evaluable/Missing | 12
  Aspergillus Syndromes (A. flavus): number analyzed (Participants) | 2
  Aspergillus Syndromes (A. flavus): Success | 1
  Aspergillus Syndromes (A. flavus): Failure | 1
  Aspergillus Syndromes (A. flavus): Not Evaluable/Missing | 0
  Aspergillus Syndromes (other): number analyzed (Participants) | 14
  Aspergillus Syndromes (other): Success | 2
  Aspergillus Syndromes (other): Failure | 7
  Aspergillus Syndromes (other): Not Evaluable/Missing | 5

10. Secondary Outcome: Percentage of Participants With a Mycological Response by Fungal Disease
Description: The percentage of participants with a Mycological Response as determined by the DRC by fungal disease, at disease specific timepoints. Mycological Response: evidence of eradication or clearance of cultures or reduction of fungal burden, as assessed by a quantitative and validated laboratory marker.
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Mycological response was evaluated based on culture, microscopy and other biomarkers of fungal infection.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Acute Invasive Candidiasis, including Candidemia: number analyzed (Participants) | 61
  Acute Invasive Candidiasis, including Candidemia: Success | 16
  Acute Invasive Candidiasis, including Candidemia: Failure | 10
  Acute Invasive Candidiasis, including Candidemia: Not Evaluable/Missing | 35
  Chronic Invasive Candidiasis: number analyzed (Participants) | 43
  Chronic Invasive Candidiasis: Success | 4
  Chronic Invasive Candidiasis: Failure | 4
  Chronic Invasive Candidiasis: Not Evaluable/Missing | 35
  Esophageal Candidiasis: number analyzed (Participants) | 16
  Esophageal Candidiasis: Success | 2
  Esophageal Candidiasis: Failure | 5
  Esophageal Candidiasis: Not Evaluable/Missing | 9
  Oropharyngeal Candidiasis: number analyzed (Participants) | 14
  Oropharyngeal Candidiasis: Success | 7
  Oropharyngeal Candidiasis: Failure | 4
  Oropharyngeal Candidiasis: Not Evaluable/Missing | 3
  Chronic Mucocutaneous Candidiasis: number analyzed (Participants) | 13
  Chronic Mucocutaneous Candidiasis: Success | 6
  Chronic Mucocutaneous Candidiasis: Failure | 6
  Chronic Mucocutaneous Candidiasis: Not Evaluable/Missing | 1
  Vulvovaginal Candidiasis: number analyzed (Participants) | 32
  Vulvovaginal Candidiasis: Success | 11
  Vulvovaginal Candidiasis: Failure | 13
  Vulvovaginal Candidiasis: Not Evaluable/Missing | 8
  Disseminated/Invasive Dimorphic Fungi: number analyzed (Participants) | 3
  Disseminated/Invasive Dimorphic Fungi: Success | 0
  Disseminated/Invasive Dimorphic Fungi: Failure | 1
  Disseminated/Invasive Dimorphic Fungi: Not Evaluable/Missing | 2
  Chronic Pulmonary Aspergillosis: number analyzed (Participants) | 6
  Chronic Pulmonary Aspergillosis: Success | 1
  Chronic Pulmonary Aspergillosis: Failure | 4
  Chronic Pulmonary Aspergillosis: Not Evaluable/Missing | 1
  Allergic Bronchopulmonary Aspergillosis: number analyzed (Participants) | 5
  Allergic Bronchopulmonary Aspergillosis: Success | 1
  Allergic Bronchopulmonary Aspergillosis: Failure | 2
  Allergic Bronchopulmonary Aspergillosis: Not Evaluable/Missing | 2
  Invasive Pulmonary Aspergillosis: number analyzed (Participants) | 29
  Invasive Pulmonary Aspergillosis: Success | 3
  Invasive Pulmonary Aspergillosis: Failure | 7
  Invasive Pulmonary Aspergillosis: Not Evaluable/Missing | 19
  Other Emerging Fungi: number analyzed (Participants) | 11
  Other Emerging Fungi: Success | 2
  Other Emerging Fungi: Failure | 2
  Other Emerging Fungi: Not Evaluable/Missing | 7

11. Secondary Outcome: Percentage of Participants With a Mycological Response by Enrollment Category
Description: The percentage of participants with a Mycological Response as determined by the DRC by enrollment category, at disease specific timepoints. Mycological Response: evidence of eradication or clearance of cultures or reduction of fungal burden, as assessed by a quantitative and validated laboratory marker.
  Disease specific timepoints: End of Treatment (EoT) for invasive candidiasis, EoT or Day 84 for Chronic Mucocutaneous Candidiasis, Test of Cure (TOC) for Vulvovaginal Candidiasis, EoT or Day 90 for Chronic Pulmonary Aspergillosis, EoT or Day 90 Allergic Bronchopulmonary Aspergillosis and EoT for all other diseases. Mycological response was evaluated based on culture, microscopy and other biomarkers of fungal infection.
Time Frame: as for outcome 1
Population: Intent to Treat (ITT) includes all participants enrolled in the study who received at lease one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Refractory: number analyzed (Participants) | 128
  Refractory: Success | 21
  Refractory: Failure | 33
  Refractory: Not Evaluable/Failure | 74
  Resistence: number analyzed (Participants) | 134
  Resistence: Success | 28
  Resistence: Failure | 19
  Resistence: Not Evaluable/Failure | 87
  Intolerance: number analyzed (Participants) | 29
  Intolerance: Success | 7
  Intolerance: Failure | 10
  Intolerance: Not Evaluable/Failure | 12
  Toxicities: number analyzed (Participants) | 17
  Toxicities: Success | 1
  Toxicities: Failure | 5
  Toxicities: Not Evaluable/Failure | 11
  Relapse: number analyzed (Participants) | 18
  Relapse: Success | 5
  Relapse: Failure | 2
  Relapse: Not Evaluable/Failure | 11

12. Secondary Outcome: Percentage of Participants With a Recurrence of Baseline Fungal Disease
Description: The percentage of participants with a recurrence of their baseline fungal disease as assessed by the DRC at the 25-Day Follow Up (FU) for Vulvovaginal Candidiasis and at the 6-Week FU for all other diseases as assessed by the DRC. Recurrence is defined as having Global Response at end of treatment or test of cure, but re-emergence of the baseline fungal disease during the post treatment follow-up. Re-emergence is required to be with the same species and involving the same site identified at baseline.
Time Frame: 42 days for vulvovaginal candidiasis and 6 weeks after End of Treatment (up to 180 days after treatment start) for all other diseases.
Population: Intent to Treat (ITT) population (any participant who was enrolled in the study and received at least one dose of study drug) that achieved a Global Response.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Acute Invasive Candidiasis including Candidemia: number analyzed (Participants) | 40
  Acute Invasive Candidiasis including Candidemia: Recurrence | 0
  Acute Invasive Candidiasis including Candidemia: No Recurrence | 35
  Acute Invasive Candidiasis including Candidemia: Not Evaluable | 5
  Chronic Invasive Candidasis: number analyzed (Participants) | 30
  Chronic Invasive Candidasis: Recurrence | 0
  Chronic Invasive Candidasis: No Recurrence | 29
  Chronic Invasive Candidasis: Not Evaluable | 1
  Candidemia only: number analyzed (Participants) | 13
  Candidemia only: Recurrence | 0
  Candidemia only: No Recurrence | 11
  Candidemia only: Not Evaluable | 2
  Esophageal Candidiasis: number analyzed (Participants) | 9
  Esophageal Candidiasis: Recurrence | 3
  Esophageal Candidiasis: No Recurrence | 5
  Esophageal Candidiasis: Not Evaluable | 1
  Oropharyngeal Candidiasis: number analyzed (Participants) | 9
  Oropharyngeal Candidiasis: Recurrence | 2
  Oropharyngeal Candidiasis: No Recurrence | 7
  Oropharyngeal Candidiasis: Not Evaluable | 0
  Chronic Mucotaneous Candidiasis: number analyzed (Participants) | 7
  Chronic Mucotaneous Candidiasis: Recurrence | 4
  Chronic Mucotaneous Candidiasis: No Recurrence | 2
  Chronic Mucotaneous Candidiasis: Not Evaluable | 1
  Vulvovaginal Candidiasis: number analyzed (Participants) | 28
  Vulvovaginal Candidiasis: Recurrence | 6
  Vulvovaginal Candidiasis: No Recurrence | 18
  Vulvovaginal Candidiasis: Not Evaluable | 4
  Disseminated/Invasive Dimorphic Fungi: number analyzed (Participants) | 1
  Disseminated/Invasive Dimorphic Fungi: Recurrence | 1
  Disseminated/Invasive Dimorphic Fungi: No Recurrence | 0
  Disseminated/Invasive Dimorphic Fungi: Not Evaluable | 0
  Chronic Pulmonary Aspergillosis: number analyzed (Participants) | 1
  Chronic Pulmonary Aspergillosis: Recurrence | 0
  Chronic Pulmonary Aspergillosis: No Recurrence | 1
  Chronic Pulmonary Aspergillosis: Not Evaluable | 0
  Allergic Bronchopulmonary Aspergillosis: number analyzed (Participants) | 0
  Allergic Bronchopulmonary Aspergillosis: Recurrence | 0
  Allergic Bronchopulmonary Aspergillosis: No Recurrence | 0
  Allergic Bronchopulmonary Aspergillosis: Not Evaluable | 0
  Invasive Pulmonary Aspergillosis: number analyzed (Participants) | 12
  Invasive Pulmonary Aspergillosis: Recurrence | 2
  Invasive Pulmonary Aspergillosis: No Recurrence | 10
  Invasive Pulmonary Aspergillosis: Not Evaluable | 0
  Other: number analyzed (Participants) | 7
  Other: Recurrence | 0
  Other: No Recurrence | 6
  Other: Not Evaluable | 1

13. Secondary Outcome: Percentage of Participants Surviving at Day 30 or Day 42
Description: Percentage of participants with invasive candidiasis surviving at Day 30 post-Baseline or percentage of participants with other fungal diseases surviving at Day 42 post-Baseline.
Time Frame: Day 30 post-Baseline for Invasive Candidiasis and Day 42 post-Baseline for all other fungal diseases.
Population: Intent to Treat (ITT) Population - any participant enrolled in the study who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Participants
  Acute Invasive Candidiasis: number analyzed (Participants) | 41
  Acute Invasive Candidiasis: Alive | 39
  Acute Invasive Candidiasis: Dead | 1
  Acute Invasive Candidiasis: Unknown | 1
  Chronic Invasive Candidiasis: number analyzed (Participants) | 43
  Chronic Invasive Candidiasis: Alive | 43
  Chronic Invasive Candidiasis: Dead | 0
  Chronic Invasive Candidiasis: Unknown | 0
  Candidemia: number analyzed (Participants) | 20
  Candidemia: Alive | 17
  Candidemia: Dead | 1
  Candidemia: Unknown | 2
  Esophageal Candidiasis: number analyzed (Participants) | 16
  Esophageal Candidiasis: Alive | 15
  Esophageal Candidiasis: Dead | 0
  Esophageal Candidiasis: Unknown | 1
  Oropharyngeal Candidiasis: number analyzed (Participants) | 14
  Oropharyngeal Candidiasis: Alive | 14
  Oropharyngeal Candidiasis: Dead | 0
  Oropharyngeal Candidiasis: Unknown | 0
  Chronic Mucocutaneous Candidiasis: number analyzed (Participants) | 13
  Chronic Mucocutaneous Candidiasis: Alive | 13
  Chronic Mucocutaneous Candidiasis: Dead | 0
  Chronic Mucocutaneous Candidiasis: Unknown | 0
  Vulvovaginal Candidiasis: number analyzed (Participants) | 32
  Vulvovaginal Candidiasis: Alive | 32
  Vulvovaginal Candidiasis: Dead | 0
  Vulvovaginal Candidiasis: Unknown | 0
  Disseminated/Invasive Dimorphic Fungi: number analyzed (Participants) | 3
  Disseminated/Invasive Dimorphic Fungi: Alive | 3
  Disseminated/Invasive Dimorphic Fungi: Dead | 0
  Disseminated/Invasive Dimorphic Fungi: Unknown | 0
  Chronic Pulmonary Aspergillosis: number analyzed (Participants) | 6
  Chronic Pulmonary Aspergillosis: Alive | 5
  Chronic Pulmonary Aspergillosis: Dead | 0
  Chronic Pulmonary Aspergillosis: Unknown | 1
  Allergic Bronchopulmonary Aspergillosis: number analyzed (Participants) | 5
  Allergic Bronchopulmonary Aspergillosis: Alive | 5
  Allergic Bronchopulmonary Aspergillosis: Dead | 0
  Allergic Bronchopulmonary Aspergillosis: Unknown | 0
  Invasive Pulmonary Aspergillosis: number analyzed (Participants) | 29
  Invasive Pulmonary Aspergillosis: Alive | 22
  Invasive Pulmonary Aspergillosis: Dead | 6
  Invasive Pulmonary Aspergillosis: Unknown | 1
  Other Emerging Fungi: number analyzed (Participants) | 11
  Other Emerging Fungi: Alive | 10
  Other Emerging Fungi: Dead | 0
  Other Emerging Fungi: Unknown | 1

14. Secondary Outcome: Time to Death From Any Cause
Description: Time to death from any cause in days per Fungal Disease
Time Frame: Six weeks after End of Treatment (EOT). EOT for Vulvovaginal Candidiasis is Day 7, Chronic Mucocutaneous Candidiasis is up to Day 84, Chronic Pulmonary Aspergillus and Allergic Bronchopulmonary Aspergillosis is up to Day 90 and up to Day 180 for other.
Population: Safety Population - All subjects who received at least one dose of study drug and who had at least one safety assessment post-Baseline.
Measure: Median (95% Confidence Interval); unit: Number of days
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
Number of days
  Acute Invasive Candidiasis: number analyzed (Participants) | 41
  Acute Invasive Candidiasis | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Candidemia: number analyzed (Participants) | 20
  Candidemia | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Chronic Invasive Candidiasis: number analyzed (Participants) | 43
  Chronic Invasive Candidiasis | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Vulvovaginal Candidiasis: number analyzed (Participants) | 32
  Vulvovaginal Candidiasis | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Esophageal Candidiasis: number analyzed (Participants) | 16
  Esophageal Candidiasis | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Oropharyngeal Candidiasis: number analyzed (Participants) | 14
  Oropharyngeal Candidiasis | NA [122 to NA] — Not Evaluable: Insufficient number of participants with events
  Chronic Mucocutaneous Candidiasis: number analyzed (Participants) | 13
  Chronic Mucocutaneous Candidiasis | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Diffuse/Invasive Dimorphic Fungi: number analyzed (Participants) | 3
  Diffuse/Invasive Dimorphic Fungi | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Chronic Pulmonary Aspergillosis: number analyzed (Participants) | 6
  Chronic Pulmonary Aspergillosis | NA [125 to NA] — Not Evaluable: Insufficient number of participants with events
  Allergic Bronchopulmonary Aspergillosis: number analyzed (Participants) | 5
  Allergic Bronchopulmonary Aspergillosis | NA [NA to NA] — Not Evaluable: Insufficient number of participants with events
  Invasive Pulmonary Aspergillosis: number analyzed (Participants) | 29
  Invasive Pulmonary Aspergillosis | 282 [282 to NA] — Not Evaluable: Insufficient number of participants with events
  Other Emerging Fungi: number analyzed (Participants) | 11
  Other Emerging Fungi | 270 [270 to NA] — Not Evaluable: Insufficient number of participants with events

15. Secondary Outcome: Describe Ibrexafungerp Plasma Concentrations
Description: Ibrexafungerp plasma concentrations measured at specified timepoints prior to and after administration of study drug for participants that received the following dose regimen:
  Day 1 and 2 loading dose - 750mg BID Day 3 onwards - 750mg QD
Time Frame: Day 2 post-dose, Day 3-5 pre-dose, Dat 7-10 pre-dose.
Population: Pharmacokinetic (Pk) Population - all enrolled participants who provided at least one Pk sample and with no deviations significant enough to affect interpretation of the Pk data.
Measure: Median (Full Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Ibrexafungerp (SCY-078)
Number analyzed (Participants) | 233
nanograms per milliliter (ng/mL)
  Day 2 post-dose: number analyzed (Participants) | 74
  Day 2 post-dose | 479 [0 to 1790]
  Day 3-5 pre-dose: number analyzed (Participants) | 127
  Day 3-5 pre-dose | 644 [9.21 to 1980]
  Day 7-10 pre-dose: number analyzed (Participants) | 119
  Day 7-10 pre-dose | 571 [0 to 1810]

ADVERSE EVENTS:
Time Frame: Six weeks after End of Treatment (EOT). EOT for Vulvovaginal Candidiasis is Day 7, Chronic Mucocutaneous Candidiasis is up to Day 84, Chronic Pulmonary Aspergillus and Allergic Bronchopulmonary Aspergillosis is up to Day 90 and up to Day 180 for other.
Arm/Group | Ibrexafungerp (SCY-078)
All-Cause Mortality (participants affected / at risk) | 15/233
Serious Adverse Events (participants affected / at risk) | 102/233
Other Adverse Events (participants affected / at risk) | 215/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrexafungerp (SCY-078) (N=233)
Abdominal abscess (Infections and infestations) | 1 (1)
Abdominal infection (Infections and infestations) | 2 (2)
Abscess (Infections and infestations) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (8)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Acute lymphocytic leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2)
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Blastic plasmacytoid dendritic cell neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (2)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5)
Cystitis (Infections and infestations) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (6)
Device dislocation (Product Issues) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Disease progression (General disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Drug clearance decreased (Investigations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 2 (2)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1)
General physical health deterioration (General disorders) | 1 (3)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
HCoV-NL63 infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcaemic seizure (Nervous system disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Kidney rupture (Injury, poisoning and procedural complications) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (2)
Liver abscess (Infections and infestations) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Septic shock (Infections and infestations) | 4 (4)
Shock (Vascular disorders) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Stenotrophomonas bacteraemia (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (7)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Venoocclusive disease (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp (SCY-078) (N=233)
Diarrhoea (Gastrointestinal disorders) | 163
Nausea (Gastrointestinal disorders) | 111
Vomiting (Gastrointestinal disorders) | 92
Abdominal Pain (Gastrointestinal disorders) | 26
Abdominal Pain Upper (Gastrointestinal disorders) | 18
Urinary Tract Infection (Infections and infestations) | 22
COVID-19 (Infections and infestations) | 14
Pyrexia (General disorders) | 31
Fatigue (General disorders) | 20
Headache (Nervous system disorders) | 38
Dizziness (Nervous system disorders) | 17
Decreased Appetite (Metabolism and nutrition disorders) | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 13
Acute Kidney Injury (Renal and urinary disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03059992/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03059992/SAP_001.pdf